CLINICAL TRIAL: NCT06420700
Title: A Multi-site, Prospective Registry of Patients Undergoing Combined Gastric Mucosal Ablation With Endoscopic Sleeve Gastroplasty at True You Weight Loss
Brief Title: Ablation Registry (Combined Gastric Mucosal Ablation With Endoscopic Sleeve Gastroplasty for Weight Loss)
Status: Recruiting | Type: Observational
Sponsor: True You Weight Loss (Other)
Responsible Party: Sponsor
Other Study IDs: RGT-001
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: ghrelin; fundus ablation; gastric mucosal ablation; endoscopic sleeve gastroplasty; ESG-MAX; obesity; ablation; hunger; True You Weight Loss
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — (Optional) Gastric fundus biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined gastric mucosal ablation with endoscopic sleeve gastroplasty: All patients included in the multi-site, prospective registry will undergo the combined gastric mucosal ablation with endoscopic sleeve gastroplasty procedure, regardless of their participation in the research study.
  Interventions: Procedure: Combined gastric mucosal ablation with endoscopic sleeve gastroplasty

INTERVENTIONS:
Procedure: Combined gastric mucosal ablation with endoscopic sleeve gastroplasty — Combined gastric mucosal ablation with endoscopic sleeve gastroplasty in the treatment of adults with obesity

SUMMARY:
The purpose of this study is to construct a multi-site, prospective registry to evaluate the clinical outcomes of patients who have undergone combined gastric mucosal ablation with endoscopic sleeve gastroplasty at True You Weight Loss.

DETAILED DESCRIPTION:
Obesity is a chronic disease state driven by the imbalance of caloric intake and expenditure and mediated by multiple central and peripheral pathways that may serve as targets for therapeutic interventions. The endoscopic sleeve gastroplasty (ESG) is a per oral gastric remodeling technique that employs full-thickness suturing to imbricate the stomach along the greater curvature to achieve a restricted, sleeve-like configuration. While the ESG recapitulates the configuration of a gastric sleeve, it has not yet been shown to achieve as robust weight loss outcomes compared to the laparoscopic sleeve gastrectomy (LSG). A major difference between ESG and LSG is that the former does not involve the gastric fundus. The proximal stomach, and the fundus in particular, produces ghrelin, the only known orexigenic hormone, which has been linked to increased calorie intake and weight gain. Studies have observed reduced levels of ghrelin along multiple timepoints following LSG and this has been attributed to targeting of the fundus, as bariatric surgeries that did not involve the fundus did not see a decrease in circulating plasma ghrelin. In contrast, in a small comparative study of ESG and LSG, patients who had undergone ESG did not show any decrease in fasting ghrelin levels, ostensibly due to fundic-sparing. In a preliminary, first-in-human study conducted by True You Weight Loss (ABLATE Weight), gastric fundus ablation via hybrid argon plasma coagulation was followed sequentially by ESG after 6 months. In this 10-patient study, fundus ablation was performed safely in all cases and without serious adverse events. A subsequent first-in-human study (ABLATE WEIGHT 2) further investigated gastric fundus ablation in a single-stage approach by combining fundus ablation and ESG during the same endoscopic session. Preliminary data revealed enhanced clinical effectiveness for the single-stage approach when compared to traditional endoscopic sleeve gastroplasty while maintaining a clinically feasible safety profile. By constructing a multi-site, prospective registry, the investigators aim to longitudinally collect and assess the clinical outcomes and characteristics of patients undergoing combined gastric mucosal ablation with endoscopic sleeve gastroplasty (ESG) at True You Weight Loss.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 65 years old
2. BMI ≥ 28 and ≤55 kg/m²
3. Willingness to comply with the substantial lifelong dietary restrictions required by the procedure.
4. Ability to give informed consent
5. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.
6. Those who plan to receive the gastric mucosal ablation with ESG procedure at True You Weight Loss regardless of the research

Exclusion Criteria:

1. Patients that do not meet eligibility requirements for the study as per the Principal Investigator's standard selection criteria
2. Active psychological issues preventing participation in a life-style modification program as determined by a psychologist.
3. Patients who are pregnant or breast-feeding.
4. Patients currently taking weight-loss medications or other therapies for weight loss within the prior 6 months.
5. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating.
6. At the discretion of the PI for subject safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (Age ≥ 18 years and ≤ 65 and BMI ≥ 28 and ≤55 kg/m²) who underwent combined gastric mucosal ablation with endoscopic sleeve gastroplasty at True You Weight Loss locations (Cary, NC and Atlanta, GA) regardless of their voluntary participation in the research
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Total Body Weight Loss (TBWL) from Baseline | 12 Months
  Measured percent change in total body weight over time following combined Gastric Mucosal Ablation. %TBWL = (pre-op weight - post op body weight) / (pre-op weight) * 100 measured as a percentage.

SECONDARY OUTCOMES:
Percent Change in Total Body Weight Loss (TBWL) from Baseline | 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 24 Months
  Measured percent change in total body weight over time following combined Gastric Mucosal Ablation. %TBWL = (pre-op weight - post op body weight) / (pre-op weight) * 100 measured as a percentage.
Percent Excess Weight Loss from Baseline (EWL) | 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 24 Months
  Measured excess weight loss percentage from baseline following combined Gastric Mucosal Ablation. %EWL = (pre-op weight - post op body weight) / (pre-op weight - ideal body weight) * 100
  Ideal Body Weight (IBW):
  Males: IBW = 50 kg + 2.3 kg for each inch over 5 feet Females: IBW = 45.5 kg + 2.3 kg for each inch over 5 feet
Change in Body Mass Index (BMI) from Baseline | 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 24 Months
  Measured Body Mass Index (BMI) from baseline following combined Gastric Mucosal Ablation. Body Mass Index (BMI) = (Weight in kilograms) / ((Height in meters)^2)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - True You Weight Loss, Atlanta, Georgia
  - True You Weight Loss, Cary, North Carolina

REFERENCES:
- [Background] Fukunishi Y. [Electron microscopic findings in peripheral nerve lesions of nude mouse inoculated with M. leprae--perineural lesion]. Nihon Rai Gakkai Zasshi. 1985 Jul-Sep;54(3):82-7. doi: 10.5025/hansen1977.54.82. No abstract available. Japanese. PMID 3915747
- [Background] Cummings DE, Overduin J. Gastrointestinal regulation of food intake. J Clin Invest. 2007 Jan;117(1):13-23. doi: 10.1172/JCI30227. PMID 17200702
- [Background] Goitein D, Lederfein D, Tzioni R, Berkenstadt H, Venturero M, Rubin M. Mapping of ghrelin gene expression and cell distribution in the stomach of morbidly obese patients--a possible guide for efficient sleeve gastrectomy construction. Obes Surg. 2012 Apr;22(4):617-22. doi: 10.1007/s11695-011-0585-9. PMID 22231739
- [Background] Anderson B, Switzer NJ, Almamar A, Shi X, Birch DW, Karmali S. The impact of laparoscopic sleeve gastrectomy on plasma ghrelin levels: a systematic review. Obes Surg. 2013 Sep;23(9):1476-80. doi: 10.1007/s11695-013-0999-7. PMID 23794092
- [Background] McCarty TR, Jirapinyo P, Thompson CC. Effect of Sleeve Gastrectomy on Ghrelin, GLP-1, PYY, and GIP Gut Hormones: A Systematic Review and Meta-analysis. Ann Surg. 2020 Jul;272(1):72-80. doi: 10.1097/SLA.0000000000003614. PMID 31592891
- [Background] Langer FB, Reza Hoda MA, Bohdjalian A, Felberbauer FX, Zacherl J, Wenzl E, Schindler K, Luger A, Ludvik B, Prager G. Sleeve gastrectomy and gastric banding: effects on plasma ghrelin levels. Obes Surg. 2005 Aug;15(7):1024-9. doi: 10.1381/0960892054621125. PMID 16105401
- [Background] Peterli R, Wolnerhanssen B, Peters T, Devaux N, Kern B, Christoffel-Courtin C, Drewe J, von Flue M, Beglinger C. Improvement in glucose metabolism after bariatric surgery: comparison of laparoscopic Roux-en-Y gastric bypass and laparoscopic sleeve gastrectomy: a prospective randomized trial. Ann Surg. 2009 Aug;250(2):234-41. doi: 10.1097/SLA.0b013e3181ae32e3. PMID 19638921
- [Background] Lopez-Nava G, Negi A, Bautista-Castano I, Rubio MA, Asokkumar R. Gut and Metabolic Hormones Changes After Endoscopic Sleeve Gastroplasty (ESG) Vs. Laparoscopic Sleeve Gastrectomy (LSG). Obes Surg. 2020 Jul;30(7):2642-2651. doi: 10.1007/s11695-020-04541-0. PMID 32193741
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503